CLINICAL TRIAL: NCT05247567
Title: Quaternary Ammonium and Immunization in Hairdressers
Acronym: AQTIFF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: there is not enough volounteer for the trial
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP211212; 2021-A01722-39 (Other: ID-RCB)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Quaternary Ammonium; Hypersensitivity
Keywords: hypersensitivity; hairdressers; quaternary ammonium
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First year students (Other): Students in their first year of Hairdressing School
  Interventions: Biological: serum punction; Biological: skin swab in elbow folds
- Third year students (Other): Students in their third year of Hairdressing School
  Interventions: Biological: serum punction; Biological: skin swab in elbow folds

INTERVENTIONS:
Biological: serum punction — A blood sample inclusion and at the end of study visit
Biological: skin swab in elbow folds — passage of a cotton swab in the crease of the elbow at the inclusion

SUMMARY:
"Quaternary ammonium ions (QA) are surfactants and microbicide products found in a large number of household products, disinfectants and cosmetics.

Professional exposure to QA causes allergic diseases of the skin and lung (asthma). It is also the firs cause of occupational rhinitis since 2000.

Several studies have found a link between exposure to some disinfectants and asthma in specific population. Moreover, a study showed that exposure to QA found in hairdressing products could also be a risk factor to allergy to neuro-muscular blocking agents.

However, the prevalence of QA sensitization amongst hairdressers is not known, sensitization mechanisms have been poorly characterized. To date, there is no recommendation regarding QA exposure nor classification of QA by toxicity. Finally, the link between hairdressing QA and drug allergy have not been confirmed yet.

The investigator hypothesize that it is possible to sensitize to QA by exposure to hairdressing products and then to declare allergic diseases. The investigator plan to study this hypothesis in an observational prospective cohort of hairdressing students by measuring both sensitization markers in blood and QA exposure. "

DETAILED DESCRIPTION:
Quaternary ammonium ions (QA) are surfactants and microbicide products found in a large number of household products, disinfectants and cosmetics.

Professional exposure to QA causes allergic diseases of the skin and lung (asthma). It is also the first cause of occupational rhinitis since 2000.

Several studies have found a link between exposure to some disinfectants and asthma in specific population. The responsibility of the QA in asthma can be demonstrated by in vivo testing (inhalation challenge). Some QA have been shown to directly activate the immune system, in particular didecyldimethylammonium chloride, a common disinfectant, that was demonstrated to act as a sensitizer.

Neuromuscular blocking agents (NMBA) are drugs used during surgery to relax muscles. They all have QA moieties and can trigger sometimes severe IgE-mediated allergic reaction (anaphylaxis). The epitope of these drugs recognized by the Immunoglobulin E (IgE) antibodies are precisely the QA moieties. However, the origin of these IgE is unknown as a significant proportion of patients have anaphylaxis on the first exposure an NMBA. A study showed that exposure to QA found in hairdressing products was linked to anti-IgE QA and then might also be a risk factor to allergy to NMBA.

Thus, QA exposure is strongly suspected to be linked to allergic diseases. However, the prevalence of QA sensitization amongst hairdressers is not known, sensitization mechanisms have been poorly characterized. To date, there is no recommendation regarding QA exposure nor classification of QA by toxicity. Finally, the link between hairdressing QA and drug allergy have not been confirmed yet.

We hypothesize that it is possible to sensitize to QA by exposure to hairdressing products and then to declare allergic diseases. We plan to study this hypothesis in an observational prospective cohort of hairdressing students by measuring both sensitization markers in blood and QA exposure.

The investigator will study 2 groups of hairdressing students :

* first year students, before the beginning of their apprenticeship in a Salon
* third year students Both groups will be programmed for a visit in the Center for Clinical Investigation of the Bichat Hospital, Paris, France. During this visit, after obtention of written consent, a blood sample (10 mL) will be collected in a serum collection tube, and a form about exposure to QA will be filled by the student.

For first year students only, a similar visit will be planned at the end of their studies (2 years after inclusion) Serum will be collected and frozen in a biobank in Bichat Hospital. Total and QA specific IgE and Immunoglobulin G (IgG) will be measured.

Differences in prevalence will be assessed by Fischer's exact test, the link between exposure levels and IgG and IgE levels will be assessed by Spearman correlation, and the evolution of IgE and IgG concentrations over time will be measured by a paired hypothesis test chosen according to data's distribution."

ELIGIBILITY:
Inclusion criteria :

* Being at least 16
* Being regularly registered in a Hairdressing school in first and second year
* Mastery of French language

Exclusion criteria :

* No French speaking parents for underage students
* People under legal guardianship
* French special Health Insurance for non-residents (AME)"

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Difference between prevalence of quaternary ammonium sensitization between first and third year hairdressing students | 1 day
  Sensitization will be evaluated as the percentage of students with serum anti-Quaternary Ammonium IgE concentration >0,35 KU/L

SECONDARY OUTCOMES:
Comparison of quaternary ammonium sensitization of hairdresser to a age-matched birth cohort | 1 day
  The difference in prevalence of quaternary ammonium sensitization (seric IgE>0,35 kU/L) between the first year students and a reference population of the same age and geographic origin
Evaluation of the link between quaternary ammonium sensitization and other measured biological parameters and clinical data collected | 1 day
  Measure of the correlation between all collected parameters and concentrations of anti-quaternary ammonium concentrations
the relative variation of IgE anti-quaternary ammonium concentrations of first year students at inclusion and after two years of study | 2 years
the relative variation of IgG anti-quaternary ammonium concentrations of first year students at inclusion and after two years of study | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luc de Chaisemartin, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided